CLINICAL TRIAL: NCT06501690
Title: Feasibility of a Bedtime Variability Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Emily Hohman, Associate Research Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00025204
Record Dates: First submitted 2024-07-02; First posted 2024-07-15 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Sleep
Keywords: sleep; bedtime

STUDY DESIGN:
Intervention Model Description: Participants will complete 3, one week long intervention periods in a randomized order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Habitual bedtime (No Intervention): For one week, children will follow their habitual bedtime.
- Late bedtime (Experimental): For one week, children will go to bed one hour later than their habitual bedtime
  Interventions: Behavioral: Late bedtime
- Variable bedtime (Experimental): For one week, children will go to bed at a prescribed time that will vary each day within +/- 1 hour of habitual bedtime.
  Interventions: Behavioral: Variable bedtime

INTERVENTIONS:
Behavioral: Late bedtime — Participants will go to bed 1 hour later than their habitual bedtime
  Arms: Late bedtime
Behavioral: Variable bedtime — Participants will go to bed at a prescribed time that varies each day within +/-1 hour of habitual bedtime
  Arms: Variable bedtime

SUMMARY:
The purpose of this study is to find out if parents and children 6-10 years old are willing and able to follow a protocol to be used to study the effects of short and/or variable sleep in children. During each of three, one-week long periods, parents will have their child follow one of the following bedtime schedules: 1) habitual bedtime; 2) 1 hour later bedtime; or 3) variable bedtime (+/- 1 hour of habitual bedtime each day). Children will wear a sleep tracker and parents will complete daily diaries. Participants will answer questions about their experiences completing the protocol.

DETAILED DESCRIPTION:
The purpose of this study is to find out if parents and children 6-10 years old are willing and able to follow a protocol to be used to study the effects of short and/or variable sleep in children. Children with medical conditions or taking medications affecting sleep, or children who do not have a regular bedtime, will be excluded. During each of three, one-week long periods, parents will have their child follow one of the following bedtime schedules: 1) habitual bedtime; 2) 1 hour later bedtime; or 3) variable bedtime (+/- 1 hour of habitual bedtime each day). Children will wear a sleep tracker and parents will complete daily diaries. Participants will answer questions about their experiences completing the protocol. Participants will attend an initial enrollment visit to complete consent and receive instruction on the protocol. Participants will then complete the three experimental conditions in a randomized, counterbalanced order. Participants will complete a phone or Zoom check in at the end of the first two conditions, and an in-person or Zoom visit at the end of the third condition where their opinions about the protocol feasibility and acceptability will be assessed, answer any questions, and provide them instruction for the next condition (when applicable).

ELIGIBILITY:
Inclusion Criteria:

* Child age 6-10 years
* Parent age 18 years or older
* Child has a regular bedtime (goes to bed within 30 minutes of the same time on 5 or more days per week)

Exclusion Criteria:

* Child has a medical condition impacting sleep (e.g., narcolepsy, sleep apnea)
* Child has a developmental disorder or delay (e.g., autism, Down syndrome)
* Child regularly takes supplements or medications (prescription or over the counter) for sleep, such as melatonin or antihistamines
* Not English speaking
* Not willing to follow bedtime protocol
* Residing in the same household as a current or previous participant (i.e., only 1 child per household may complete study)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to bedtime protocol | Daily during each of the 3, one-week intervention periods
  Parents will report on the time their child went to bed

SECONDARY OUTCOMES:
Parent perception of feasibility of following the protocol (semi-structured interview) | At the end of 3 week study
  Parents will provide qualitative answers to questions about their perceptions of following the protocol, including but not limited to whether the protocol was easy to follow, disruptive to their life, disruptive to their child's life.
Sleep duration | Daily during each of the 3, one-week intervention period
  Child sleep duration during each intervention period, measured by actigraphy

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No